CLINICAL TRIAL: NCT04407975
Title: Effect of Single Dose Antenatal Betamethasone on the Incidence of Neonatal Respiratory Morbidity After Elective Cesarean Section at Term: A Prospective Double Blinded Placebo Controlled Trial
Brief Title: Effect of Single Dose Antenatal Betamethasone on Neonatal Respiratory Morbidity After Elective Cesarean
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Manal Hubeish, Principal Investigator, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 642020
Record Dates: First submitted 2020-05-18; First posted 2020-05-29 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Morbidity
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betamethasone (Experimental): Patients will receive 14 mg (2 ml) intramuscular betamethasone
  Interventions: Other: Betamethasone
- Placebo (Placebo Comparator): Patients will receive an equivalent volume of normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Betamethasone — A single injection will be administered to the patient at least 24 hours before undergoing C-section. This injection will be prepared in the hospital's pharmacy to contain betamethasone
  Arms: Betamethasone
Other: Placebo — A single injection will be administered to the patient. This injection will be prepared in the hospital's pharmacy to contain normal saline.
  Arms: Placebo

SUMMARY:
Patients undergoing elective C-section will be randomized into two groups. The first group will receive one dose of Betamethasone at least 24 hours before scheduled C-section. The second group will receive placebo.

DETAILED DESCRIPTION:
This is a prospective double blinded randomized clinical trial. Patients will be randomized into two groups. Group A will receive one dose of Betamethasone at least 24 hours before scheduled C-section. Group B will receive placebo. The maternal and neonatal outcomes will be studied in order to assess the effect of Betamethasone on respiratory morbidity of the newborn infant.

ELIGIBILITY:
Inclusion Criteria:

* women with singleton or multiple gestation,
* between 37 and 40 weeks of pregnancy (as calculated from the first day of the last menstrual period)

Exclusion Criteria:

* any medical problem that could affect fetal well-being;
* evidence of intrauterine infection,
* oligohydramnios,
* fetal congenital malformations,
* preeclampsia,
* maternal hypertension,
* severe fetal rhesus sensitization,
* antepartum hemorrhage,
* Intrauterine growth restriction
* preterm rupture of membranes
* preterm delivery
* previously received antenatal steroids less than one month ago
* those who decline to participate in the study.

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with respiratory morbidity | at birth
  Neonatal respiratory morbidity will be assessed through oxygen saturation, Apgar score and Silverman score

SECONDARY OUTCOMES:
Admission to Neonatal Intensive Care Unit (NICU) | up to 2 weeks
  Reasons for NICU admission and length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hubeish, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon